CLINICAL TRIAL: NCT00026143
Title: Phase II Trial of Interleukin-12 (NSC #672423, IND #6798) Followed by Interferon Alfa-2B in Patients With Metastatic Malignant Melanoma
Brief Title: Interleukin-12 and Interferon Alfa in Treating Patients With Metastatic Malignant Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02816; CALGB-500001; CDR0000068990; U10CA031946 (NIH)
Record Dates: First submitted 2001-11-09; First posted 2003-01-27 (Estimated); Last update posted 2013-06-05 (Estimated); Status verified 2013-06

CONDITIONS: Recurrent Melanoma; Stage IV Melanoma
MeSH Terms: conditions — Melanoma | interventions — Interleukin-12 Subunit p35; Interleukin-12; Interferon-alpha; Interferon Alfa-n3; Introns; Interferon alpha-2

ARMS (1):
- Arm I (Experimental): Patients receive interleukin-12 IV over 5-15 seconds on day 1 and interferon alfa subcutaneously on days 2-6. Treatment repeats every 2 weeks in the absence of unacceptable toxicity. Patients are reassessed after 6 courses. Patients with a complete response receive 2 additional courses. Patients with a partial response or stable disease continue treatment in the absence of disease progression.
  Interventions: Biological: recombinant interleukin-12; Biological: recombinant interferon alfa; Other: laboratory biomarker analysis

INTERVENTIONS:
Biological: recombinant interleukin-12 — Given IV
  Other Names: cytotoxic lymphocyte maturation factor; IL-12; interleukin-12; natural killer cell stimulatory factor; Ro 24-7472
Biological: recombinant interferon alfa — Given SC
  Other Names: Alferon N; alpha interferon; IFN-A; Intron A; Roferon-A
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
Phase II trial to study the effectiveness of combining interleukin-12 and interferon alfa in treating patients who have metastatic malignant melanoma. Interleukin-12 may kill tumor cells by stopping blood flow to the tumor and by stimulating a person's white blood cells to kill cancer cells. Interferon alfa may interfere with the growth of the cancer cells. Combining interleukin-12 and interferon alfa may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the clinical response rates in patients with metastatic malignant melanoma treated with rhIL-12 and interferon alfa-2b.

II. To estimate the progression-free survival in patients with metastatic malignant melanoma treated with rhIL-12 and interferon alfa-2b.

SECONDARY OBJECTIVES:

I. To measure serum levels of interferon-gamma. II. To measure levels of JAK-STAT signaling intermediates in patient PBMCs and tumor samples.

III. To analyze interferon-alpha-induced STAT signaling in patient PBMCs. IV. To determine the expression of IFN-regulated genes in patient PBMCs and tumor tissues.

V. To determine the pattern of gene expression induced by treatment with IL-12 and interferon-alpha using DNA microarray techniques in patient PBMCs.

OUTLINE: This is a multicenter study.

Patients receive interleukin-12 IV over 5-15 seconds on day 1 and interferon alfa subcutaneously on days 2-6. Treatment repeats every 2 weeks in the absence of unacceptable toxicity. Patients are reassessed after 6 courses. Patients with a complete response receive 2 additional courses. Patients with a partial response or stable disease continue treatment in the absence of disease progression.

Patients are followed every 3 months for 1 year and then every 6 months for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological diagnosis of cutaneous melanoma and clinical evidence of distant, metastatic, non-resectable regional lymphatic, or extensive in transit recurrent disease
* Patients must have measurable disease; measurable disease is defined as the presence of at least one measurable lesion; if the measurable disease is restricted to a solitary lesion, its neoplastic nature should be confirmed by cytology/histology; measurable lesions are defined as lesions that can be accurately measured in at least one dimension with the longest diameter >= 20 mm using conventional techniques or >= 10 mm with spiral CT scan

  * Lesions that are considered intrinsically non-measurable include the following:

    * Bone lesions;
    * Leptomeningeal disease;
    * Ascites;
    * Pleural/pericardial effusion;
    * Inflammatory breast disease;
    * Lymphangitis cutis/pulmonis;
    * Abdominal masses that are not confirmed and followed by imaging techniques;
    * Lytic lesions;
    * Lesions that are situated in a previously irradiated area
* No history of peripheral neuropathy, brain metastases or other central nervous system disease
* No history of/active autoimmune disease, hemolytic anemia or concurrent requirement for corticosteroids, including topical or inhaled
* No hepatitis BSAg, known HIV disease or other major active illness; patients with risk factors for HIV should be tested; patients with these illnesses are more likely to experience significant side effects from the study treatment
* No history of severe peptic ulcer disease or gastrointestinal bleeding unless there is objective evidence that the condition is inactive or resolved
* No uncontrolled or severe cardiovascular disease, diabetes, pulmonary disease, or infection
* No chemotherapy, radiotherapy, or anti-hormonal therapy within three weeks prior to the initiation of therapy on this study
* No prior therapy with IL-12
* No prior therapy with IFN-alpha for metastatic disease (e.g., biochemotherapy); prior adjuvant therapy with IFN-a is acceptable as long as the patient remained disease-free for 12 months or longer following the last IFN-a treatment
* No prior cytokine therapy for metastatic disease (e.g., high-dose IL-2)
* No more than one prior chemotherapy regimen
* CTC (ECOG) performance status 0-1
* Non-pregnant, non-nursing; treatment under this protocol would expose an unborn child to significant risks; women and men of reproductive potential should agree to use an effective means of birth control; women of child-bearing age will undergo pregnancy testing
* ANC >= 1500/μL
* Platelets >= 100,000/μL
* Hemoglobin > 9 g/dL (may be post transfusion or may receive EPO)
* U-HCG or Serum HCG Negative (if patient of child-bearing potential)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2001-10; Primary Completion 2004-07 (Actual)

PRIMARY OUTCOMES:
Response rate | Up to 2 years
PFS | From registration until time of documented progression of disease or death from any cause, assessed up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: William Carson, Principal Investigator — Cancer and Leukemia Group B
Locations (1):
- Cancer and Leukemia Group B, Chicago, Illinois, United States